CLINICAL TRIAL: NCT04243889
Title: Fetoscopic Spina Bifida Repair Using a Cryopreserved Human Umbilical Cord Allograft (NEOX Cord 1K®) as a Meningeal Patch
Brief Title: Fetoscopic NEOX Cord 1K® Spina Bifida Repair
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Ramesha Papanna, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-19-1051
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Spina Bifida; Myelomeningocele; Myeloschisis
Keywords: Neox Cord 1K; Fetoscopic repair; Cryopreserved human umbilical cord
MeSH Terms: conditions — Spinal Dysraphism; Meningomyelocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- NEOX Cord 1K applied fetoscopically (Experimental): Patients intending to undergo open in-utero spina bifida repair, will be offered to be screened for an alternative minimally invasive approach. All eligible pregnant mothers' fetuses within the trial will receive NEOX Cord 1K® as a spinal cord cover to close the developmental defect. In some cases, at the discretion of the Neurosurgeon, NEOX Cord 1K® may be required to cover the skin. All eligible subjects meeting all inclusion criteria but none of the exclusion criteria may be enrolled.
  Interventions: Device: NEOX Cord 1K

INTERVENTIONS:
Device: NEOX Cord 1K — Under general anesthesia and tocolysis, in-utero repair begins with a laparotomy that is followed by exteriorization of the uterus. The fetus is then positioned by external cephalic version. Uterine entry will be accessed using 3 cannulas, followed by heated-humidified carbon dioxide insufflation for visualization. Then, fetoscopically the placode will be examined and dissected. The lesion will be repaired using NEOX Cord 1K® (HUC) for closure of the first layer over the neural placode. Primary closure of the skin will then occur, or NEOX Cord 1K® (HUC) will be used for skin closure at the discretion of the neurosurgeon. Finally, the laparotomy site will be sutured in multiple layers.

SUMMARY:
To fetoscopically use cryopreserved human umbilical cord allografts, named NEOX Cord 1K®, as a spinal cord cover of spina bifida defects. This procedure will be performed to create a watertight seal covering over the spinal cord in order to decrease the incidence rates of postnatal morbidities. For larger skin defects, NEOX Cord 1K® may be used as a skin cover.

ELIGIBILITY:
Inclusion Criteria:

Maternal inclusion criteria:

* Singleton pregnancy
* Gestational age at screening is 19 to 25 5/7 weeks and gestational age at surgery is 22 to 25 6/7 weeks
* Maternal age: 18 years and older
* Body mass index < 40 kg/m2
* No preterm birth risk factors (short cervix, history of previous preterm delivery)
* No previous uterine incision in the active uterine segment
* Willing to undergo an open fetal repair if the fetoscopic approach is unsuccessful

Fetal inclusion criteria:

* Spina bifida defect between T1 to S1 vertebral levels
* Chiari II malformation
* No evidence of kyphosis (curved spine)
* No major life-threatening fetal anomaly unrelated to spina bifida
* Normal karyotype, or normal Chromosomal microarray analysis (CMA), or a CMA with variants of unknown significance

Exclusion Criteria:

Maternal exclusion criteria:

* Non-resident of the United States
* Multifetal pregnancy
* Poorly controlled insulin-dependent pregestational diabetes
* Poorly controlled A2 diabetes mellitus (A2DM) insulin-dependent diabetes
* Current or planned cerclage or documented history of an incompetent cervix
* Placenta previa or placental abruption
* Short cervix of < 20 mm
* Obesity as defined by a body mass index of > 40 kg/m2
* Previous spontaneous singleton delivery prior to 37 weeks
* Maternal-fetal Rh isoimmunization, Kell sensitization, or a history of neonatal alloimmune thrombocytopenia
* HIV or Hepatitis-B positive status
* Known Hepatitis-C positivity
* Uterine anomaly such as large or multiple fibroids or a mullerian duct abnormality that is diagnosed via imaging prior to surgery, which that are unavoidable during surgery
* Other medical conditions which are contraindication to surgery or general anesthesia
* Patient does not have a support person
* Inability to comply with the travel and follow-up requirements of the trial
* Patient does not meet psychosocial standardized assessment criteria
* Participation in this or another intervention study that influences maternal and fetal morbidity and mortality
* Maternal hypertension
* Zika virus positivity
* Allergy/history of drug reaction to Amphotericin B

Fetal exclusion criteria:

* Major fetal anomaly not related to spina bifida
* Kyphosis in the fetus of 30 degrees or more
* Ventriculomegaly greater than 15 mm and no movements noted at hip and knee joints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2029-03-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with successful fetoscopic repair of the defect using NEOX Cord 1K® | Immediately after repair procedure
  A digital image of the fetal repair site will be captured during and immediately after the repair. The images will be sent to three independent blinded neurosurgeons for review of successful closure of the defect. More than best of three votes will be considered as the result.

SECONDARY OUTCOMES:
Number of patients with intact repair of the defect, defined as no cerebrospinal fluid leakage and no dehiscence at the repair site. | Birth
Number of patients with intact repair of the defect as defined as no cerebrospinal fluid leakage and no dehiscence at the repair site. | 12 months ± 2 months

OTHER OUTCOMES:
Assessment of Arnold-Chiari malformation II | birth discharge or 1 month + 30 days, 12 ± 2 months, and 60-66 months post birth
  Assessment of Arnold-Chiari malformation II as measured by MRI of head
Number of patients with absence of brain stem kinking as assessed by MRI evaluation. | birth-discharge or 1 month + 30 days, 12 ± 2 months, and 60-66 months post birth
Number of patients with lower extremity motor and sensory levels exceeding the anatomical level of the lesion by ≥ 2 segments. | 2 ± 2 months, 30-36 months and 60-66 months post birth
Number of patients who can ambulate with or without the use of orthotics or devices. | 12 ± 2 months, 30-36 months and 60-66 months post birth
Number of patients with no spinal cord tethering as assessed by a lumbar spine MRI. | birth-discharge or 1 month + 30 days, 12 ± 2 months, and 60-66 months post birth
Number of patients with absence of syringomyelia as assessed by an MRI. | 12 ± 2 months post birth
Number of patient with the absence of an epidermoid cyst at the repair site, determined by MRI. | birth-discharge or 1 month + 30 days, 12 ± 2 months, and 60-66 months post birth
Number of patients needing de-tethering surgery before the 12 month ± 2 month visit as clinically indicated. | 12 ± 2 months
Developmental motor scales as assessed by the Bayley IV test. | 30-36 months follow up post birth
Adaptive behavior as assessed by the Vineland Adaptive Behavior Scales III | 30-36 months and 60-66 months post delivery
Achievement as measured by the Woodcock-Johnson IV Test of Achievement test | 60-66 months post birth
Assess brain stem function, as measured by the child's swallowing profile | 12 ± 2 months; 30-36 months and 60-66 months post birth
Urodynamic function assessments | 12 ± 2 months, 30-36 months and 60-66 months post birth
  Objective measures of the function of the lower urinary tract by evaluating post-void residual urine
Bowel function assessments bowel movements. | 12 ± 2 months, 30-36 months and 60-66 months post birth
  Bowel function as assessed by observation of neurogenic bowel incontinence or constipation
Verbal and non-verbal intelligence as measured by the Kaufman Brief Intelligence Test 2 (KBIT-2) | 60-66 months post delivery
Manual dexterity and bimanual coordination as determined by the Purdue Pegboard test | 60-66 months post delivery
Executive function testing as measured by the Behavior Rating Inventory of Executive Function 2 (BRIEF2) test | 60-66 months post delivery
Visual motor integration as assessed by the Beery Visual-Motor Integration test | 60-66 months post delivery
Quality of Life as assessed by the Parkin Spina Bifida Health-Related Quality of Life questionnaire | 60-66 months post delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ramesha Papanna, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Backley S, Bergh EP, Garnett J, Li R, Maroufy V, Jain R, Fletcher S, Tsao K, Austin M, Johnson A, Papanna R. Fetal cardiovascular changes during open and fetoscopic in-utero spina bifida closure. Ultrasound Obstet Gynecol. 2024 Aug;64(2):193-202. doi: 10.1002/uog.27579. PMID 38207160